CLINICAL TRIAL: NCT02258685
Title: Factors Mediating Gut Microbiota Dysbiosis and Metabolic Disease in HIV Patients.
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 14-1595
Record Dates: First submitted 2014-10-01; First posted 2014-10-07 (Estimated); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: HIV; Lipodystrophy
Keywords: Gut microbiota composition
MeSH Terms: conditions — Lipodystrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood and rectosigmoid biopsy tissue will be collected.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Cohort A1: ART-treated HIV-infected individuals with lipodystrophy
- Cohort A2: ART-treated HIV-infected individuals without lipodystrophy
- Cohort A3: HIV-1 infected individuals naïve to ART
- Cohort A4: HIV-1 seronegative individuals who are at a high risk for infection
- Cohort B1: A subset of subjects from Cohort A: ART-treated HIV-infected individuals with HIV-associated dysbiosis
- Cohort B2: A subset of subjects from Cohort A: ART-treated HIV-infected individuals without HIV-associated dysbiosis

SUMMARY:
This study plans to learn more about immune responses in intestinal (gut) tissue in people with human immunodeficiency virus (HIV) infection. This study will determine whether change in the composition of gut bacteria in HIV infected individuals is related to a high prevalence of chronic gut inflammation and metabolic disease. The investigators will also investigate immune-modulatory properties of specific bacteria that correlate with disease both by characterizing which functional genes are selected for in their genomes and by stimulating immune cells isolated from blood and gut tissue with bacterial isolates. This work will establish whether gain/loss of bacterial drivers/suppressors of information in the gut contributes to metabolic disease in HIV-infected individuals.

DETAILED DESCRIPTION:
This is a prospective cohort and cross-sectional case-control study. Study participation will last up to 2 months and 93 participants will be enrolled. Participants will be evaluated for lipodystrophy, asked to complete food & gastrointestinal symptoms questionnaires and provide stool samples. A subset of participants will be asked to have a flexible sigmoidoscopy (mucosal biopsy).

Cohort A will consist of 93 participants:

Cohort A1: ART (Antiretroviral therapy) -treated HIV-infected individuals with lipodystrophy (n=35) Cohort A2: ART-treated HIV-infected individuals without lipodystrophy (n=18) Cohort A3: HIV-1 infected individuals naïve to ART (n=20) Cohort A4: HIV-1 seronegative individuals who are at a high risk for infection (n=20)

Cohort B will be a selected subset of subjects from Cohort A:

Cohort B1: ART-treated HIV-infected individuals with HIV-associated dysbiosis (n=10) Cohort B2: ART-treated HIV-infected individuals without HIV-associated dysbiosis (n=10)

ELIGIBILITY:
Inclusion Criteria:

* Men and women; 18 years to 65 years (All Cohorts)
* Subjects with chronic HIV-1 Infection defined as a positive ELISA confirmed by a positive Western Blot or plasma HIV-1 RNA level >1,000 copies/mL at any time in the past. (Cohorts A1, A2 & A3)
* HIV-1 seronegative (Cohort A4)
* Either with or without lipodystrophy (to be assessed at Visit 1)
* Body mass index (BMI) between 21-29 mg/kg2 and weight stable for at least 3 months (All Cohorts)
* Antiretroviral therapy (ART) naïve (Cohort A3): <10 days of ART treatment at any time prior to Visit 1 or previously on ART but off treatment for the previous 6 months prior to Visit 1
* Long-term ART (Cohort A1 & A2): Must be on same antiretroviral treatment and have a plasma HIV-1 RNA <25 copies/mL for 3-6 months prior to Visit 1.Liver function tests not greater than 2x normal, normal kidney and thyroid function. Fasting glucose must be <110 mg/dl
* Liver function tests not greater than 2x normal, normal kidney and thyroid function. Fasting glucose must be <110 mg/dl
* ART-treated individuals whose microbiota resembles those with untreated HIV infection and ART-treated individuals whose microbiota resembles the HIV-negative control cohort (equal numbers with and without lipodystrophy).(Cohort B; a subset of Cohort A)

Exclusion Criteria:

* Gastrointestinal disease such as inflammatory bowel disease, Clostridium difficile colitis or celiac sprue.
* history of bowel resection, bleeding disorder, history of hyperglycemia, treated with high-dose glucocorticoid therapy or alpha-interferon in past year Current use of anticoagulant therapy
* Daily use of aspirin or nonsteroidal antiinflammatory drugs (NSAIDs) with inability to withhold drug for 7 days before and after a rectosigmoid biopsy procedure.
* Used antibiotics within the prior three months
* Pregnancy
* Current use of proton pump inhibitors and H2-blockers
* Active opportunistic or other chronic infection, such as hepatitis B or C or an active malignancy
* Patient inability to participate in the study, such as inability to undergo venipuncture, completion of questionnaire or mucosal biopsy (if selected) procedures that form part of the inclusion/exclusion criteria or part of the outcome measure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV positive and HIV negative subjects (with and without lipodystrophy) between 18 and 65 years old.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Determine the gut microbiota composition using 16S ribosomal RNA (rRNA) sequencing of fecal samples | 2 months
  Compare the gut microbiota composition of HIV-positive subjects with and without lipodystrophy and long-term ART, and HIV-negative controls with diet and metabolic and immune activation markers in blood.
Determine of gut microbiota composition using rectosigmoid biopsy tissue | 2 months
  Compare the gut microbiota composition of HIV-positive ART-treated individuals by CD4+ populations and immune activation markers in gut-associated lymphoid tissues (GALT)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Lozupone, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States